CLINICAL TRIAL: NCT01572896
Title: An Internet-based Self-management Program for Adolescents With Arthritis: A Randomized Controlled Trial
Brief Title: An Internet-based Self-management Program for Adolescents With Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinician Scientist, Clinical Nurse Specialist/NP, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000028028
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Juvenile Idiopathic
Keywords: adoloescent; internet self-management; managing JIA
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taking Charge Experimental Group (Experimental)
  Interventions: Behavioral: Taking Charge: Managing JIA Online
- Control Group (Active Comparator)
  Interventions: Behavioral: Standard Medical Care and JIA Resource Center

INTERVENTIONS:
Behavioral: Taking Charge: Managing JIA Online — In addition to standard medical care, adolescents in the experimental group will receive the "Taking Charge: Managing JIA Online" Internet self-management program. The intervention is a 12-module interactive multi-component treatment protocol - that consists of JIA-specific education, self-management strategies, and social support - that is available in English and French.
  Arms: Taking Charge Experimental Group
Behavioral: Standard Medical Care and JIA Resource Center — The control group is designed to control for the potential effects on outcomes of time, attention and computer use during the intervention and through the 9-month follow-up period. In addition to standard medical care, adolescents in the attention control group will be provided with access to a self-guided patient education study website, which will have two components: basic patient educational materials about JIA ("JIA Resource Centre") and online assessments.
  Arms: Control Group

SUMMARY:
The purpose of this study is to demonstrate the effectiveness of the "Taking Charge: Managing JIA Online" Internet intervention, when compared with an attention (static education only websites) control group in improving pain and HRQL as well as other health outcomes (anxiety, depression, treatment adherence, pain coping, knowledge, and self-efficacy) in adolescents with JIA. The proposed study will enroll and randomize 294 adolescents with JIA attending 10 pediatric rheumatology hospital clinics in the Canada to either the experimental or control groups.

DETAILED DESCRIPTION:
In summary, no rigorous Internet self-management intervention has been undertaken to improve HRQL, symptoms, treatment adherence, knowledge, and self-efficacy in youth with JIA. The proposed "Managing JIA Online" Trial will rigorously examine the effects of this Internet intervention on HRQL and other health outcomes thereby filling a significant gap in our knowledge related to promotion of self-management care for adolescents with JIA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 and ≤ 18 years.
* Diagnosed with JIA (using International League of Associations for Rheumatology classification criteria)83 by their rheumatologist.
* Adolescents and parent/ primary caregiver are able to speak and read either English or French.
* Participants are willing and able to complete online measures. There will be no restrictions on medication use for this study.

Exclusion Criteria:

* Cognitive impairments (as assessed by reviewing medical chart and consultation with the patient's rheumatologist)
* Major co-morbid illnesses which may mitigate HRQL assessment

  * Excluded medical illnesses: inflammatory bowel disease, fibromyalgia, cancer, genetic disorders, diabetes
  * Excluded psychiatric conditions: post-traumatic stress disorder, panic disorder, bipolar disorder, psychosis, depression and major mood disorders. Adolescents currently on medications for major depression, bipolar disorder or psychosis would also be excluded.
* Adolescents that are currently participating in other CBT interventions.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 333 (Actual)
Dates: Start 2012-04; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Pain | 12 months
  Pain will be measured using the Recalled Pain Inventory - Short Form.91 The RPI measures current as well as least, average and worst pain intensity, pain unpleasantness, and pain interference ratings over the past week with items rated on a 11-point numerical rating scale (NRS) (e.g., 0 = 'no pain' to 10 = 'severe pain') and painful body locations. This 11-item measure has evidence of construct validity
Health-related Quality of Life (HRQL) | Baseline
  HRQL will be measured using the teen and parent PedsQL Rheumatology Modules.13 Both of the PedsQL rheumatology modules contain a 22-item self-report and parent scale with five subscales: pain and hurt, daily activities, treatment, worry, and communication.
Pain | Baseline
  Pain will be measured using the Recalled Pain Inventory - Short Form.91 The RPI measures current as well as least, average and worst pain intensity, pain unpleasantness, and pain interference ratings over the past week with items rated on a 11-point numerical rating scale (NRS) (e.g., 0 = 'no pain' to 10 = 'severe pain') and painful body locations. This 11-item measure has evidence of construct validity
Pain | 3months
  Pain will be measured using the Recalled Pain Inventory - Short Form.91 The RPI measures current as well as least, average and worst pain intensity, pain unpleasantness, and pain interference ratings over the past week with items rated on a 11-point numerical rating scale (NRS) (e.g., 0 = 'no pain' to 10 = 'severe pain') and painful body locations. This 11-item measure has evidence of construct validity
Health-related Quality of Life (HRQL) | 6 months
  HRQL will be measured using the teen and parent PedsQL Rheumatology Modules.13 Both of the PedsQL rheumatology modules contain a 22-item self-report and parent scale with five subscales: pain and hurt, daily activities, treatment, worry, and communication.
Pain | 6 months
  Pain will be measured using the Recalled Pain Inventory - Short Form.91 The RPI measures current as well as least, average and worst pain intensity, pain unpleasantness, and pain interference ratings over the past week with items rated on a 11-point numerical rating scale (NRS) (e.g., 0 = 'no pain' to 10 = 'severe pain') and painful body locations. This 11-item measure has evidence of construct validity
Health-related Quality of Life (HRQL) | 3 months
  HRQL will be measured using the teen and parent PedsQL Rheumatology Modules.13 Both of the PedsQL rheumatology modules contain a 22-item self-report and parent scale with five subscales: pain and hurt, daily activities, treatment, worry, and communication.
Health-related Quality of Life (HRQL) | 12 months
  HRQL will be measured using the teen and parent PedsQL Rheumatology Modules.13 Both of the PedsQL rheumatology modules contain a 22-item self-report and parent scale with five subscales: pain and hurt, daily activities, treatment, worry, and communication.

SECONDARY OUTCOMES:
Emotional Symptoms | Baseline, 3 months, 6 months and 12 months post-intervention
  Anxiety and depression will each be assessed using two, separate 8-item PROMIS (Patient Reported Outcomes Measurement Information System) scales.
Adherence | Baseline, 3 months, 6 months and 12 months post-intervention
  Adherence to medical treatment will be assessed using the 34-item Child Adherence Report Questionnaire (CARQ)
Pain Coping | Baseline, 3 months, 6 months and 12 months post-intervention
  Pain coping will be measured using the 18-item Pain Coping Questionnaire106, which is an internationally used measure of pain coping strategies in the pediatric population and has been validated in youth with arthritis.
Juvenile Idiopathic Arthritis (JIA) | Baseline, 3 months, 6 months and 12 months post-intervention
  JIA-specific knowledge will be measured using 9-items from the Medical Issues, Exercise, Pain and Social Support Questionnaire (MEPS).
Self-Efficacy | Baseline, 3 months, 6 months and 12 months post-intervention
  Self-efficacy will be measured using the Children's Arthritis Self-Efficacy (CASE) scale which is an 11-item measure.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Stinson, RN, PhD, CPNP, Principal Investigator — The Hospital for Sick Children
Locations (11):
- Canada (11):
  - Hamilton Health Sciences, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Alberta Children's Hospital, Calgary
  - Stollery Children's Hospital, Edmonton
  - IWK Health Centre, Halifax
  - Montreal Children's Hospital, Montreal
  - Children's Hospital of Eastern Ontario, Ottawa
  - Royal University, Saskatoon
  - Janeway Children's Health and Rehabilitation Centre, St. Johns
  - BC Children's Hospital, Vancouver
  - Winnepeg Children's Hospital, Winnepeg

REFERENCES:
- [Derived] Stinson JN, Lalloo C, Hundert AS, Campillo S, Cellucci T, Dancey P, Duffy C, Ellsworth J, Feldman BM, Huber AM, Johnson N, Jong G, Oen K, Rosenberg AM, Shiff NJ, Spiegel L, Tse SML, Tucker L, Victor JC. Teens Taking Charge: A Randomized Controlled Trial of a Web-Based Self-Management Program With Telephone Support for Adolescents With Juvenile Idiopathic Arthritis. J Med Internet Res. 2020 Jul 29;22(7):e16234. doi: 10.2196/16234. PMID 32723728